CLINICAL TRIAL: NCT06973902
Title: Advanced Heart Failure: The Predictive Value of Dobutamine Echo-stress in the Clinical Response to Cardiac Contractility Modulation Therapy (CCM)
Brief Title: The Predictive Value of Dobutamine Echo-stress in the Clinical Response to CCM Therapy in Advanced HF
Acronym: PREDICT-CCM
Status: Recruiting | Type: Observational
Sponsor: Quovadis Associazione (Other)
Collaborators: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: PREDICT-CCM
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Symptomatic Congestive Heart Failure
Keywords: Heart failure; systolic left ventricular dysfunction; low-dose dobutamine stress echocardiography; Cardiac Contractility Modulation (CCM)
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- DeltaESV>=15%: Subjects showing a reduction of 15% or more in LVESV through pre-implant low-dose dobutamine echocardiography stress testing
  Interventions: Device: Cardiac Contractility Modulation (CCM) implant
- DeltaESV<15%: Subjects showing a reduction of less than 15% in LVESV through pre-implant low-dose dobutamine echocardiography stress testing
  Interventions: Device: Cardiac Contractility Modulation (CCM) implant

INTERVENTIONS:
Device: Cardiac Contractility Modulation (CCM) implant — Subjects participating in the study carry or will carry the Cardiac Contractility Modulation (CCM) medical device "OPTIMIZER Smart Mini" by Impulse Dynamics (USA). It is indicated for use in patients over 18 years of age with symptomatic heart failure due to systolic left ventricular dysfunction, despite appropriate medical treatment.
  The OPTIMIZER Smart Mini Implantable Pulse Generator is a programmable device with an internal battery and telemetry functions.
  The OPTIMIZER Smart Mini is connected to two or three implantable leads, two of which are implanted in the right ventricle and one, optionally, in the right atrium.

SUMMARY:
The goal of this observational cohort study, which is both retrospective and prospective, is to evaluate the long-term clinical and instrumental response to Cardiac Contractility Modulation (CCM) treatment in adult subjects suffering from symptomatic heart failure (HF) due to systolic left ventricular dysfunction, despite adequate medical therapy. Based on the response to stress echocardiography with preimplantation low-dose Dobutamine, the main questions it aims to answer are:

* What is the proportion of subjects who experience a clinical response to CCM therapy at 12 months (NYHA reduction ≥ 1 class)?
* There was a reduction in the number of hospitalizations, visits to the Emergency Department, and access to day hospital facilities for more than 4 hours compared to the year before the study (e.g., by intravenous infusion of cardiac inotropic drugs)?
* What is the estimated change in the quality-of-life score using the "Quality of Life Questionnaire with Heart Failure - Minnesota" (MLHFQ) between baseline and the end of follow-up?
* What is the change in walking distance between baseline and the end of the follow-up in the walk test (6MWT) (optional)?
* What is the difference in NT-proBNP levels between baseline and the end of follow-up? Participants are already receiving CCM support as part of their regular medical care for heart failure.

DETAILED DESCRIPTION:
-Introductory summary When no other therapeutic options are available, CCM can be a helpful complement to treating heart failure, improving quality of life, and prolonging survival. Still, the high cost and availability of implants in qualified centers limit their use.

Then, searching for indicators that maximize the benefit/risk ratio is appropriate. According to the study's proponents, the contractile reserve of the left ventricle assessed by stress echo to low-dose Dobutamine may be among the most promising indicators for this purpose.

Introduction Heart failure (H.F.) has a very poor prognosis in terms of mortality, quality of life, and functional capacity. It is one of the most important cardiovascular diseases in terms of global prevalence and healthcare costs. Despite appropriate medical care, many patients experience frequent hospitalizations and limitations in daily activities (1).

The prevalence of heart failure ranges between 1% and 3% in the general adult population in industrialized countries. It is expected to increase substantially due to the availability of better diagnostic tools and medical treatments that prolong life after diagnosis of HF (2).

The latest international guidelines on the management of reduced ejection fraction H.F. recommend a timely approach with the simultaneous introduction of the four main categories of drugs (ACE inhibitors or ARNIs, beta-blockers, mineralocorticoid receptor antagonists (MRAs), and SGLT2 inhibitors). If drug therapy alone is not sufficient or not well tolerated by the subject, or if there is a disorder in the conduction of the electrical impulse (in particular, a left bundle branch block), it is possible to associate it with electrical therapy, which consists of the implantation of biventricular cardiac devices (pacemakers or defibrillators) that resynchronize cardiac contraction (cardiac resynchronization therapy, CRT). These devices work in close synergy with anti-decompensation drugs to curb the progression of heart failure and, in some cases, restore normal cardiac contractility. Cardiac resynchronization therapy, combined with drug therapy, has been shown to improve survival and quality of life by reducing the symptoms of heart failure, increasing exercise capacity, and enabling subjects to resume many of their daily activities.

Cardiac Contractility Modulation (CCM) CRT is indicated for patients with a large QRS (>130 ms and evidence of left bundle branch block)3; however, the percentage of individuals who do not respond to CRT varies between studies, usually between 25% and 33% (4). Randomized clinical trials have shown that Cardiac Contractility Modulation (CCM) is a treatment option5 for patients with symptomatic heart failure despite optimized medical therapy and not eligible for CRT. CCM therapy has also been evaluated in patients who have not responded to CRT (6) therapy.

The implanted device for CCM consists of an implantable pulse generator (like a pacemaker) equipped with a transcutaneously rechargeable battery connected to two ventricular leads that transmit high-energy electrical impulses within the absolute refractory period of the myocardial action potential. The device has no pacing or antiarrhythmic functions and is designed to work even in patients already implanted with pacemakers or defibrillators.

The FIX-HF-47, FIX-HF-58,9, and FIX-HF-5C10 trials demonstrated the safety and efficacy of the CCM device concerning the following end-points:

* NYHA classroom improvement.
* Improvement in the quality of life (according to the Minnesota Living with Heart Failure Questionnaire - MLHFQ).
* Improvement in functional capacity at the 6-minute walk test (6MWT).
* Increased peak oxygen consumption (VO2).
* Reduction of cardiovascular death and hospitalizations for heart failure.

The CCM has been shown to improve myocardial contractility (11) by improving cardiomyocyte management of intracellular calcium. It exerts short- and long-term effects and positively modulates cardiac cell gene expression.

The Optimizer Smart system has been approved in countries where the C.E. mark applies since October 3, 2016.

The OPTIMIZER Smart System is indicated for use in patients over 18 who have symptomatic heart failure due to systolic left ventricular dysfunction despite medical and interventional therapy. CCM therapy delivered by the OPTIMIZER system has been shown to improve the clinical status, functional capacity, and quality of life and prevent hospital admissions in symptomatic patients with left heart failure who are carefully selected and followed by cardiologists experienced in the treatment of heart failure (12).

The Optimizer Smart device was FDA-approved on March 21, 2019, for delivering Cardiac Contractility Modulation (CCM) therapy. This approval is unique in that it is the first device to be granted "Breakthrough Device" status by the FDA and to have been included in the FDA's review panel for cardiovascular devices - where it received a unanimous recommendation for approval due to its favorable benefit/risk ratio and then obtained PMA approval by the FDA (12).

In the 2021 ESC guidelines for diagnosing and treating acute and chronic heart failure (13), CCM is an "under evaluation" therapy in NYHA class III/IV patients, with LVEF between 25% and 45% and QRS duration <130 ms.

In the consensus paper published in 2024 by the Heart Failure Association (HFA) and the European Heart Rhythm Association (EHRA) of the European Society of Cardiology (ESC)(14), CCM is suggested as a therapy that experienced operators who cooperate in a multidisciplinary team for heart failure should consider if symptoms persist.

It has been evaluated that, for heart failure patients with reduced ejection fraction, the addition of CCM therapy could be more convenient than OMT alone (i.e., the combined use of five classes of drugs that, individually, have already been shown to improve the prognosis of infarcted patients: acetylsalicylic acid, beta-blockers, statins, antagonists of the renin-angiotensin system, and thienopyridines), if a time horizon of the whole life is considered (15, 16).

In selected cases, and when no other therapeutic options are available, CCM can be adjunct in patients who do not respond to CRT29.

In a recent study (30), CCM significantly improved H.F. in patients with reduced ejection fraction (HFrEF), NYHA class III, and moderately prolonged QRS of 120-149 ms.

Pharmacological stress echocardiography Pharmacological stress echocardiography is indicated for the diagnosis and treatment of suspected ischemic heart disease or left ventricular dysfunction of suspected ischemic origin. The examination consists of performing an echocardiogram during the infusion of increasing drug doses that stimulate the sympathetic nervous system, stimulating the heart with an effect similar to physical exertion. The heart reacts with increased contraction force and frequency; sometimes, blood pressure can also increase. The examination helps to recognize the possible presence of stress-induced myocardial ischemia.

Other indications of stress echocardiography include quantifying contractile reserve in cardiomyopathies, evaluating cardiac valvulopathy and congenital heart disease, and evaluating diastolic function and pulmonary hypertension. The main advantages of stress echocardiography are its simplicity, low cost, wide availability, and absence of radiation (17, 18).

The most used drugs in this procedure are Dobutamine or dipyridamole. Dobutamine is a synthetic catecholamine that primarily stimulates β1 adrenergic receptors and, to a lesser extent, α1 and β2 receptors.

The protocol for standard dobutamine examination was defined in the American Society of Echocardiography (ASE) guidelines of 2007 (19). A graduated dobutamine infusion is usually administered at a 5 μg/kg starting dose per minute. The dobutamine infusion aims to achieve a heart rate of 85% of the maximum heart rate predicted for the person's age. The dose of Dobutamine is increased every 3-5 minutes to 10, 20, 30, and finally to 40 μg/kg per minute (20).

On the other hand, the "low-dose" dobutamine stress echocardiography (LDDSE) test is optimal for detecting ischemia and assessing viability by searching for the "biphasic response." A myocardial area increases its contraction at a low dose of inotropic but later becomes hypokinetic or akinetic at higher doses of dobutamine (20).

During the low-dose dobutamine stress echocardiography, the subject is stressed with Dobutamine by standardized incremental infusions of 5, 10, and 20 μg/kg/min. Each infusion dose is administered for a maximum of five minutes (18, 20, 21, 22).

As assessed by low-dose dobutamine stress echo, left ventricular contractile reserve is a helpful marker for predicting functional improvement of the left ventricle and determining long-term prognosis in patients with dilated heart disease (23).

Low-dose dobutamine stress echocardiography has proven to be a simple and effective procedure for selecting patients who are candidates for CRT, having demonstrated the correlation between contractile reserve and response to subsequent resynchronization therapy (24). The assay was also used to quantify the degree of remodeling after CRT (25) therapy.

Many CRT studies have evaluated left ventricular reverse remodeling by echocardiographic testing with low-dose Dobutamine. A positive response criterion is a reduction of left ventricular end-systolic volume (LVESV) greater than or equal to 15% (26, 27, 28).

ELIGIBILITY:
Inclusion Criteria:

* Subject of both sexes with age ≥ 18 years,
* Ability to understand and sign informed consent to participate in the study and consent to process sensitive personal data.
* Carrier of symptomatic heart failure, despite optimal medical therapy (OMT),
* Reduced left ventricular systolic function (E.F. <50%),
* It was positively evaluated for implanting a system for cardiac contractility modulation (CCM) (according to the European Society of Cardiology 2021 Guidelines on heart failure and the provisions of the C.E. mark approval)13.
* Have presented at least one hospitalization, access to the Emergency Department, or access to day hospital facilities for more than 4 hours (e.g., by intravenous infusion of cardiac inotropic drugs) in the year before implantation

Exclusion Criteria:

* Life expectancy < 1 year due to non-cardiac comorbidities that reduce prognosis,
* Presence of contraindications to the CCM implantation procedure (absence of vascular access usable for CCM implantation, active infectious processes, active severe coagulopathies, presence of mechanical tricuspid valve),
* Contraindications to the performance of the echocardiographic test under pharmacological stress (heart failure in progress, myocardial infarction in the acute phase, acute inflammatory processes of the heart muscle and/or pericardium, critical aortic valve stenosis and severe obstructions to left ventricular outflow, dissecting aneurysm of the aorta, severe arrhythmias not controlled by therapy, known hypersensitivity to the drug, intraventricular thrombi).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollable subjects who, in the participating Clinical Centers, received a CCM implant from July 1, 2024, to the start of the study will be part of the retrospective cohort, while subsequent subjects of the prospective cohort.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
New York Heart Association class variation | From enrollment to the end of follow-up, 12 months
  The proportion of subjects with clinical response to CCM therapy at 12 months, defined as a reduction of at least 1 class of the New York Heart Association Classification of the functional status of the heart (minimum value I, better outcome, and maximum value IV, worse outcome)

SECONDARY OUTCOMES:
Hospitalizations | From enrollment to the end of follow-up, 12 months
  Change in the number of hospitalizations, visits to the Emergency Department, or access to day hospital facilities for more than 4 hours (e.g., by intravenous infusion of cardiac inotropic drugs) compared to the year before the study.
Minnesota LIVING WITH HEART FAILURE Questionnaire score variation | From enrollment to the end of follow-up, 12 months
  Change in the quality-of-life score estimated with the "Minnesota LIVING WITH HEART FAILURE Questionnaire" MLHFQ (minimum value 0, better outcome, and maximum value 105, worse outcome),
6MWT variation | From enrollment to the end of follow-up, 12 months
  Change in walk distance between baseline and end of follow-up in the walk test (6MWT)
NT-proBNP variation | From enrollment to the end of follow-up, 12 months
  Change in NT-proBNP level between baseline and end of follow-up
LVESV change | From enrollment to the end of follow-up, 12 months
  The proportion of subjects with LVESV decreased by ≥ 15% on echocardiography at end-of-follow-up compared to preimplantation
VTI change | From enrollment to the end of follow-up, 12 months
  The proportion of subjects with increased integral velocity time (VTI) ≥ 20% between preimplantation and end-of-follow-up echocardiography,
LVEF change | From enrollment to the end of follow-up, 12 months
  The proportion of subjects with a 20% increase in ejection fraction (LVEF) between preimplantation and end-of-follow-up echocardiography
MR change | From enrollment to the end of follow-up, 12 months
  The proportion of subjects with progression or, conversely, improvement in Mitral Regurgitation (M.R.; classified as mild, moderate, or severe).
CRT implant | From enrollment to the end of follow-up, 12 months
  The proportion of subjects who, during follow-up, will be evolved to cardiac resynchronization system (CRT) implantation
LVAD implant | From enrollment to the end of follow-up, 12 months
  The proportion of subjects who, during follow-up, will be evolved to left ventricular assist device (LVAD) implantation,
Cardiac Transplant | From enrollment to the end of follow-up, 12 months
  The proportion of subjects who will have received a cardiac transplant during follow-up
HF death | From enrollment to the end of follow-up, 12 months
  The proportion of subjects who will die from H.F. during follow-up
AE | From enrollment to the end of follow-up, 12 months
  Rate of all procedure-related adverse events.
Re-Operation | From enrollment to the end of follow-up, 12 months
  Rate of re-operations (lead revision/replacement/infection)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zanon, MD, Study Chair — UO Cardiologia, S. Maria della Misericordia Hospital, ULSS5 Polesana, Rovigo (I)
Locations (13):
- Italy (13):
  - PO Anastasia Guerriero, Marcianise (CE), UOC Cardiologia, Marcianise, Campania
  - Clinica Montevergine, Mercogliano (AV), Laboratorio di Elettrofisiologia, Mercogliano, Campania
  - UOC Cardiologia, Osp. San Rocco, Sessa Aurunca (CE), ASL Caserta, Sessa Aurunca, Campania
  - Policlinico S.Orsola, UO Cardiologia, Bologna, Emilia-Romagna
  - OSPEDALE CASTELLI, UO Cardiologia, Anzio, Lazio
  - Elettrofisiologia e Aritmologia, ASST FBF Sacco, Milan, Lombardy
  - Fondazione Giglio, Cefalù (PA), UOC Cardiologia, Cefalù, Sicily
  - Osp. Generale Provinciale Mazzoni, UO Cardiologia, Ascoli Piceno, The Marches
  - UOC Cardiologia, Osp. Di Mirano, ULSS 3 Serenissima, Mirano, Veneto
  - UOC Cardiologia, Osp. Di Piove di Sacco (PD), ULSS 6 Euganea, Piove di Sacco, Veneto
  - UOC Cardiologia, Osp. S.Bortolo, Vicenza, ULSS 8 Berica, Vicenza, Veneto
  - UOC Cardiologia con UTIC, Osp. Di Venere, Bari
  - UO Cardiologia, S. Maria della Misericordia Hospital, ULSS5 Polesana, Rovigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rector, T., S. Kubo, and J. Cohn, Patient's self-assessment of their congestive heart failure. Part 2: content, reliability and validity of a new measure, The Minnesota Living with Heart Failure Questionnaire. Heart Failure. Heart Failure, 1987; 1:198-209
- [Background] Nagele H, Behrens S, Eisermann C. Cardiac contractility modulation in non-responders to cardiac resynchronization therapy. Europace. 2008 Dec;10(12):1375-80. doi: 10.1093/europace/eun257. Epub 2008 Sep 5. PMID 18776196
- [Background] Matsumura Y, Takata J, Kitaoka H, Hamada T, Okawa M, Kubo T, Doi Y. Low-dose dobutamine stress echocardiography predicts the improvement of left ventricular systolic function and long-term prognosis in patients with idiopathic dilated cardiomyopathy. J Med Ultrason (2001). 2006 Mar;33(1):17-22. doi: 10.1007/s10396-005-0061-z. PMID 27277614
- [Background] Pellikka PA, Nagueh SF, Elhendy AA, Kuehl CA, Sawada SG; American Society of Echocardiography. American Society of Echocardiography recommendations for performance, interpretation, and application of stress echocardiography. J Am Soc Echocardiogr. 2007 Sep;20(9):1021-41. doi: 10.1016/j.echo.2007.07.003. No abstract available. PMID 17765820
- [Background] Sicari R, Nihoyannopoulos P, Evangelista A, Kasprzak J, Lancellotti P, Poldermans D, Voigt JU, Zamorano JL; European Association of Echocardiography. Stress echocardiography expert consensus statement: European Association of Echocardiography (EAE) (a registered branch of the ESC). Eur J Echocardiogr. 2008 Jul;9(4):415-37. doi: 10.1093/ejechocard/jen175. PMID 18579481
- [Background] Narducci ML, Nurchis MC, Ballacci F, Giordano F, Calabro GE, Massetti M, Crea F, Aspromonte N, Damiani G. Cost-utility of cardiac contractility modulation in patients with heart failure with reduced ejection fraction in Italy. ESC Heart Fail. 2024 Feb;11(1):229-239. doi: 10.1002/ehf2.14538. Epub 2023 Nov 9. PMID 37943287
- [Background] Witte K, Hasenfuss G, Kloppe A, Burkhoff D, Green M, Moss J, Peel A, Mealing S, Durand Zaleski I, Cowie MR. Cost-effectiveness of a cardiac contractility modulation device in heart failure with normal QRS duration. ESC Heart Fail. 2019 Dec;6(6):1178-1187. doi: 10.1002/ehf2.12526. PMID 31997539
- [Background] Mullens W, Dauw J, Gustafsson F, Mebazaa A, Steffel J, Witte KK, Delgado V, Linde C, Vernooy K, Anker SD, Chioncel O, Milicic D, Hasenfuss G, Ponikowski P, von Bardeleben RS, Koehler F, Ruschitzka F, Damman K, Schwammenthal E, Testani JM, Zannad F, Bohm M, Cowie MR, Dickstein K, Jaarsma T, Filippatos G, Volterrani M, Thum T, Adamopoulos S, Cohen-Solal A, Moura B, Rakisheva A, Ristic A, Bayes-Genis A, Van Linthout S, Tocchetti CG, Savarese G, Skouri H, Adamo M, Amir O, Yilmaz MB, Simpson M, Tokmakova M, Gonzalez A, Piepoli M, Seferovic P, Metra M, Coats AJS, Rosano GMC. Integration of implantable device therapy in patients with heart failure. A clinical consensus statement from the Heart Failure Association (HFA) and European Heart Rhythm Association (EHRA) of the European Society of Cardiology (ESC). Eur J Heart Fail. 2024 Feb;26(2):483-501. doi: 10.1002/ejhf.3150. Epub 2024 Jan 25. PMID 38269474
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Borggrefe M, Burkhoff D. Clinical effects of cardiac contractility modulation (CCM) as a treatment for chronic heart failure. Eur J Heart Fail. 2012 Jul;14(7):703-12. doi: 10.1093/eurjhf/hfs078. Epub 2012 Jun 12. PMID 22696514
- [Background] Abraham WT, Kuck KH, Goldsmith RL, Lindenfeld J, Reddy VY, Carson PE, Mann DL, Saville B, Parise H, Chan R, Wiegn P, Hastings JL, Kaplan AJ, Edelmann F, Luthje L, Kahwash R, Tomassoni GF, Gutterman DD, Stagg A, Burkhoff D, Hasenfuss G. A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Cardiac Contractility Modulation. JACC Heart Fail. 2018 Oct;6(10):874-883. doi: 10.1016/j.jchf.2018.04.010. Epub 2018 May 10. PMID 29754812
- [Background] Abraham WT, Nademanee K, Volosin K, Krueger S, Neelagaru S, Raval N, Obel O, Weiner S, Wish M, Carson P, Ellenbogen K, Bourge R, Parides M, Chiacchierini RP, Goldsmith R, Goldstein S, Mika Y, Burkhoff D, Kadish A; FIX-HF-5 Investigators and Coordinators. Subgroup analysis of a randomized controlled trial evaluating the safety and efficacy of cardiac contractility modulation in advanced heart failure. J Card Fail. 2011 Sep;17(9):710-7. doi: 10.1016/j.cardfail.2011.05.006. Epub 2011 Jun 22. PMID 21872139
- [Background] Kadish A, Nademanee K, Volosin K, Krueger S, Neelagaru S, Raval N, Obel O, Weiner S, Wish M, Carson P, Ellenbogen K, Bourge R, Parides M, Chiacchierini RP, Goldsmith R, Goldstein S, Mika Y, Burkhoff D, Abraham WT. A randomized controlled trial evaluating the safety and efficacy of cardiac contractility modulation in advanced heart failure. Am Heart J. 2011 Feb;161(2):329-337.e1-2. doi: 10.1016/j.ahj.2010.10.025. PMID 21315216
- [Background] Borggrefe MM, Lawo T, Butter C, Schmidinger H, Lunati M, Pieske B, Misier AR, Curnis A, Bocker D, Remppis A, Kautzner J, Stuhlinger M, Leclerq C, Taborsky M, Frigerio M, Parides M, Burkhoff D, Hindricks G. Randomized, double blind study of non-excitatory, cardiac contractility modulation electrical impulses for symptomatic heart failure. Eur Heart J. 2008 Apr;29(8):1019-28. doi: 10.1093/eurheartj/ehn020. Epub 2008 Feb 12. PMID 18270213
- [Background] Campbell CM, Kahwash R, Abraham WT. Optimizer Smart in the treatment of moderate-to-severe chronic heart failure. Future Cardiol. 2020 Jan;16(1):13-25. doi: 10.2217/fca-2019-0044. Epub 2019 Dec 9. PMID 31825245
- [Background] Savarese G, Becher PM, Lund LH, Seferovic P, Rosano GMC, Coats AJS. Global burden of heart failure: a comprehensive and updated review of epidemiology. Cardiovasc Res. 2023 Jan 18;118(17):3272-3287. doi: 10.1093/cvr/cvac013. PMID 35150240
- [Background] Levy D, Kenchaiah S, Larson MG, Benjamin EJ, Kupka MJ, Ho KK, Murabito JM, Vasan RS. Long-term trends in the incidence of and survival with heart failure. N Engl J Med. 2002 Oct 31;347(18):1397-402. doi: 10.1056/NEJMoa020265. PMID 12409541

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT06973902/Prot_SAP_001.pdf